CLINICAL TRIAL: NCT03561246
Title: Incline Training to Personalize Motor Control Interventions After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N2665-R; 77797 (Other: Charleston VAMC)
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: CVA (Cerebrovascular Accident)
Keywords: Stroke; Rehabilitation; Walking; Biomechanics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Personalized training effect on SSWS and Pp - Incline (Active Comparator): Determine the efficacy of motor control deficit guided personalized training on SSWS and Paretic Propulsion (Pp).
  Incline treadmill walking: Those with a Pp <0.47 or >0.53 will undergo INCLINE training during which individuals will walk for 15 minutes at a 10-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Interventions: Other: Incline treadmill walking
- Personalized training effect on SSWS and Pp - Decline (Active Comparator): Determine the efficacy of motor control deficit guided personalized training on SSWS and Paretic Propulsion (Pp).
  Decline treadmill walking: Those with a Pp <0.47 or >0.53 will undergo DECLINE training during which individuals will walk for 15 minutes at a 10-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Interventions: Other: Decline treadmill walking
- Personalized training effect on SSWS and Pp - Level treadmill (Control) (Active Comparator): Determine the efficacy of motor control deficit guided personalized training on SSWS and Paretic Propulsion (Pp).
  Level treadmill walking: Those with a Pp <0.47 or >0.53 will undergo LEVEL training during which individuals will walk for 15 minutes at a 0-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Interventions: Other: Level Treadmill (Control)

INTERVENTIONS:
Other: Incline treadmill walking — Those with a Pp <0.47 or >0.53 will undergo INCLINE training during which individuals will walk for 15 minutes at a 10-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Arms: Personalized training effect on SSWS and Pp - Incline
Other: Decline treadmill walking — Those with a Pp <0.47 or >0.53 will undergo DECLINE training during which individuals will walk for 15 minutes at a 10-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Arms: Personalized training effect on SSWS and Pp - Decline
Other: Level Treadmill (Control) — Those with a Pp <0.47 or >0.53 will undergo LEVEL training during which individuals will walk for 15 minutes at a 0-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
  Arms: Personalized training effect on SSWS and Pp - Level treadmill (Control)

SUMMARY:
This study will evaluate the use of incline and decline treadmill training to address specific motor control deficits identified within different post-stroke walking patterns.

DETAILED DESCRIPTION:
This study seeks to develop a theory-based clinical decision-making framework for the training of walking recovery after stroke based on how different biomechanical patterns of walking illustrate distinct motor control deficits. Each participant will complete 12 sessions (three times a week for four weeks) of either INCLINE, DECLINE, or CONTROL training. Clinical and biomechanical outcome measures will be collected pre- and post-training and after a one-month follow-up period. In addition, the investigators will collect a battery of clinical outcome measures before and after training. Spatiotemporal variables (including SSWS) will be collected before and after each session. All clinical and biomechanical assessments will be conducted by an evaluator blinded to training group allocation.

ELIGIBILITY:
Inclusion Criteria:

* stroke 6 months
* residual paresis in the lower extremity (Fugl-Meyer LE motor score <34)
* ability to walk without assistance at speeds ranging from 0.2 - 1.0 m/s (with a support harness for biomechanical testing)
* Ability to walk on a treadmill without orthotic or assistive device using overhead harness system
* provision of informed consent, and 8) written approval from the primary physician (see attached sample of Medical Approval Cover Letter).

Exclusion Criteria:

* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADLs
* History of COPD or oxygen dependence
* Pre-existing neurological disorders or dementia
* History of major head trauma
* Pp between 0.47 and 0.53
* Legal blindness or severe visual impairment
* Severe arthritis or other problems that limit passive ROM
* History of DVT or pulmonary embolism within 6 months
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Cence, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - MUSC Center for Rehabilitation Research in Neurologic Conditions, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
As a clinical trial, the details of this project will be entered into ClinicalTrials.gov. Clinical data from assessment sessions will be recorded on hard copies (stored in a locked file cabinet in the Ralph H. Johnson VAMC rehabilitation research space) and entered into a RedCAP electronic database by the project coordinator immediately after each session. These data will be de-identified for further analysis. Only the PI will only have access to de-identified data. Gait data will be analyzed using a custom MATLAB program, automatically populating a LabView Data Viewer from which customized data may be retrieved. The research coordinator will check the data entry, and pool all data into a group-wide de-identified spreadsheet. All data from training sessions will also be analyzed and stored using an automated MATLAB program. All electronic data will be stored on a secure server that is backed-up nightly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completion of all study Aims. De-identified data set will be available for other investigators and registered in the NIH-supported registry.

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Training Effect on SSWS and Pp - Level Treadmill (Control): Determine the efficacy of motor control deficit guided personalized training on SSWS and Paretic Propulsion (Pp).
  Level treadmill walking: Those with a Pp <0.47 or >0.53 will undergo LEVEL treadmill training during which individuals will walk for 15 minutes at a 0-degree treadmill tilt, stopping each five minutes for monitoring of vital signs.
Period: Overall Study
Arm/Group | Personalized Training Effect on SSWS and Pp - Incline | Personalized Training Effect on SSWS and Pp - Decline | Personalized Training Effect on SSWS and Pp - Level Treadmill (Control)
Started | 19 | 19 | 17
Completed | 19 | 18 | 17
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Training Effect on SSWS and Pp - Incline | Personalized Training Effect on SSWS and Pp - Decline | Personalized Training Effect on SSWS and Pp - Level Treadmill (Control) | Total
Number analyzed (Participants) | 19 | 19 | 17 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 9 | 33
  >=65 years | 7 | 7 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.32 (8.33) | 60.79 (9.19) | 61 (10.34) | 60.96 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 4 | 17
  Male | 14 | 11 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 18 | 19 | 17 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 00 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 7 | 6 | 23
  White | 9 | 12 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 17 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed
Description: Participants will be asked to complete a 10 Meter Walk Test and a difference will be calculated between pre and post speed.
Time Frame: Pre (same day but prior to initial training session) and post (immediately following final training session) approximately 4 weeks apart.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Personalized Training Effect on SSWS and Pp - Incline | Personalized Training Effect on SSWS and Pp - Decline | Personalized Training Effect on SSWS and Pp - Level Treadmill (Control)
Number analyzed (Participants) | 19 | 18 | 17
meters/second | 0.15 (0.004) | 0.075 (0.053) | 0.127 (0.062)

2. Secondary Outcome: Change in Paretic Propulsion Symmetry
Description: Quantitative measure of the coordinated output of the paretic leg and is defined as the percentage of propulsion performed by the paretic leg.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Propulsion
Arm/Group | Personalized Training Effect on SSWS and Pp - Incline | Personalized Training Effect on SSWS and Pp - Decline | Personalized Training Effect on SSWS and Pp - Level Treadmill (Control)
Number analyzed (Participants) | 19 | 18 | 17
Percentage of Propulsion | -0.023 (0.042) | -0.034 (0.020) | 0.043 (0.013)

ADVERSE EVENTS:
Time Frame: 75 days
Description: Records were kept of non-serious adverse events in the study binder and reported to the local governing IRB in accordance with Good Clinical Practice Guidelines.
Arm/Group | Personalized Training Effect on SSWS and Pp - Incline | Personalized Training Effect on SSWS and Pp - Decline | Personalized Training Effect on SSWS and Pp - Level Treadmill (Control)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/17

LIMITATIONS AND CAVEATS:
We did not reach our target number of 60 participants due to the COVID-19 pandemic. The formatting of our study at its conclusion is different than its original presentation. Our 'arms' are updated as the incline, decline, and level treadmill conditions. We present gait speed and Pp outcomes across three conditions in our final report. We caution interpretation due to the potential impact of paretic propulsion baseline characteristic on the response to incline or decline walking conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03561246/Prot_SAP_000.pdf